CLINICAL TRIAL: NCT00119015
Title: The Addition of Montelukast to Fluticasone in the Treatment of Perennial Allergic Rhinitis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty in recruitment
Sponsor: University of Chicago (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13875B; SING-US-60-04
Record Dates: First submitted 2005-07-01; First posted 2005-07-12 (Estimated); Results first posted 2013-05-22 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-01

CONDITIONS: Rhinitis, Allergic, Perennial
Keywords: perennial allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — montelukast; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluticasone propionate + Placebo (Placebo Comparator): Fluticasone propionate nasal spray - 2 sprays in each nostril once a day for 2 weeks (200 micrograms daily)
  Placebo - 10 mg po daily for 2 weeks
  Interventions: Drug: Placebo; Drug: Fluticasone propionate
- Fluticasone propionate + Montelukast (Active Comparator): Fluticasone propionate nasal spray - 2 sprays in each nostril once a day for 2 weeks (200 micrograms daily)
  Montelukast - 10 mg po daily for 2 weeks
  Interventions: Drug: Montelukast; Drug: Fluticasone propionate

INTERVENTIONS:
Drug: Placebo
  Arms: Fluticasone propionate + Placebo
Drug: Montelukast
  Other Names: singulair
  Arms: Fluticasone propionate + Montelukast
Drug: Fluticasone propionate
  Other Names: flonase

SUMMARY:
Some people with nasal allergy symptoms continue to have symptoms even after treatment with a nasal steroid spray. The purpose of this study is to see if these patients are helped by adding another medication (montelukast) to their treatment compared to placebo (a substance that looks like the active medication but does not contain the drug).

DETAILED DESCRIPTION:
Clinicians frequently prescribe an oral H1 antihistamine for allergic rhinitis patients with residual symptoms after taking an intranasal steroid. Surprisingly, the only studies investigating this combination of drugs have failed to show added efficacy of the H1 receptor over the intranasal steroids alone. Adding montelukast, a leukotriene receptor antagonist, to an intranasal steroid has not been studied in a placebo controlled fashion. Wilson and colleagues, in an open study of patients with chronic rhinosinusitis, showed a benefit of adding montelukast.

The investigators would like to recruit perennially allergic subjects and place them on fluticasone for 2 weeks. Those subjects with residual symptoms would then be randomized to receive either placebo or montelukast in addition to continuing the fluticasone for an additional 2 weeks.

A positive study would support clinical practice and would serve as a preemptive strike against managed care plans that would not allow prescriptions for both drugs.

Hypothesis:

The addition of montelukast to treatment of a perennially allergic subject with an intranasal steroid is more effective at relieving symptoms than a placebo.

ELIGIBILITY:
Inclusion Criteria:

* A clinical history of perennial allergic rhinitis and a positive skin prick test to dust mite, cockroach, mold, or cat or dog antigens.
* Willingness of the subject to participate in and complete the study, and the ability to understand the purpose of the trial.

Exclusion Criteria:

* Physical signs or symptoms suggestive of renal, hepatic or cardiovascular disease.
* Women of childbearing potential who are pregnant, trying to become pregnant or nursing a child.
* Subjects treated with systemic steroids during the previous 30 days.
* Subjects treated with topical (inhaled, intranasal or intraocular) steroids, Nasalcrom or Opticrom during the previous 15 days.
* Subjects treated with oral antihistamines/decongestants during the previous seven days.
* Subjects treated with topical (intranasal or intraocular) antihistamines/decongestants during the previous 3 days.
* Subjects treated with immunotherapy who are escalating their dose.
* Subjects on chronic anti-asthma medications.
* Subjects with polyps in the nose or a significantly displaced septum.
* Subjects who have incurred an upper respiratory tract infection within 14 days of the start of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2005-07; Primary Completion 2008-06 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Naclerio, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Wilson AM, White PS, Gardiner Q, Nassif R, Lipworth BJ. Effects of leukotriene receptor antagonist therapy in patients with chronic rhinosinusitis in a real life rhinology clinic setting. Rhinology. 2001 Sep;39(3):142-6. PMID 11721504
- [Background] Kurowski M, Kuna P, Gorski P. Montelukast plus cetirizine in the prophylactic treatment of seasonal allergic rhinitis: influence on clinical symptoms and nasal allergic inflammation. Allergy. 2004 Mar;59(3):280-8. doi: 10.1046/j.1398-9995.2003.00416.x. PMID 14982509
- [Background] van Adelsberg J, Philip G, Pedinoff AJ, Meltzer EO, Ratner PH, Menten J, Reiss TF; Montelukast Fall Rhinitis Study Group. Montelukast improves symptoms of seasonal allergic rhinitis over a 4-week treatment period. Allergy. 2003 Dec;58(12):1268-76. doi: 10.1046/j.1398-9995.2003.00261.x. PMID 14616102
- [Background] Philip G, Nayak AS, Berger WE, Leynadier F, Vrijens F, Dass SB, Reiss TF. The effect of montelukast on rhinitis symptoms in patients with asthma and seasonal allergic rhinitis. Curr Med Res Opin. 2004 Oct;20(10):1549-58. doi: 10.1185/030079904x3348. PMID 15462688
- [Background] Di Lorenzo G, Pacor ML, Pellitteri ME, Morici G, Di Gregoli A, Lo Bianco C, Ditta V, Martinelli N, Candore G, Mansueto P, Rini GB, Corrocher R, Caruso C. Randomized placebo-controlled trial comparing fluticasone aqueous nasal spray in mono-therapy, fluticasone plus cetirizine, fluticasone plus montelukast and cetirizine plus montelukast for seasonal allergic rhinitis. Clin Exp Allergy. 2004 Feb;34(2):259-67. doi: 10.1111/j.1365-2222.2004.01877.x. PMID 14987306
- [Background] Ciprandi G, Tosca MA, Milanese M, Schenone G, Ricca V. Antihistamines added to an antileukotriene in treating seasonal allergic rhinitis: histamine and leukotriene antagonism. Eur Ann Allergy Clin Immunol. 2004 Feb;36(2):67-70, 72. PMID 15061398
- [Background] Chervinsky P, Philip G, Malice MP, Bardelas J, Nayak A, Marchal JL, van Adelsberg J, Bousquet J, Tozzi CA, Reiss TF. Montelukast for treating fall allergic rhinitis: effect of pollen exposure in 3 studies. Ann Allergy Asthma Immunol. 2004 Mar;92(3):367-73. doi: 10.1016/S1081-1206(10)61576-1. PMID 15049402
- [Background] Moinuddin R, deTineo M, Maleckar B, Naclerio RM, Baroody FM. Comparison of the combinations of fexofenadine-pseudoephedrine and loratadine-montelukast in the treatment of seasonal allergic rhinitis. Ann Allergy Asthma Immunol. 2004 Jan;92(1):73-9. doi: 10.1016/S1081-1206(10)61713-9. PMID 14756468
- [Background] Topuz B, Ogmen GG. Montelukast as an adjuvant to mainstay therapies in patients with seasonal allergic rhinitis. Clin Exp Allergy. 2003 Jun;33(6):823-6. doi: 10.1046/j.1365-2222.2003.01690.x. PMID 12801319
- [Background] Ratner PH, Howland WC 3rd, Arastu R, Philpot EE, Klein KC, Baidoo CA, Faris MA, Rickard KA. Fluticasone propionate aqueous nasal spray provided significantly greater improvement in daytime and nighttime nasal symptoms of seasonal allergic rhinitis compared with montelukast. Ann Allergy Asthma Immunol. 2003 May;90(5):536-42. doi: 10.1016/S1081-1206(10)61847-9. PMID 12775135
- [Background] Saengpanich S, deTineo M, Naclerio RM, Baroody FM. Fluticasone nasal spray and the combination of loratadine and montelukast in seasonal allergic rhinitis. Arch Otolaryngol Head Neck Surg. 2003 May;129(5):557-62. doi: 10.1001/archotol.129.5.557. PMID 12759270
- [Background] Baena-Cagnani CE, Berger WE, DuBuske LM, Gurne SE, Stryszak P, Lorber R, Danzig M. Comparative effects of desloratadine versus montelukast on asthma symptoms and use of beta 2-agonists in patients with seasonal allergic rhinitis and asthma. Int Arch Allergy Immunol. 2003 Apr;130(4):307-13. doi: 10.1159/000070218. PMID 12740532
- [Background] van Adelsberg J, Philip G, LaForce CF, Weinstein SF, Menten J, Malice MP, Reiss TF; Montelukast Spring Rhinitis Investigator Group. Randomized controlled trial evaluating the clinical benefit of montelukast for treating spring seasonal allergic rhinitis. Ann Allergy Asthma Immunol. 2003 Feb;90(2):214-22. doi: 10.1016/S1081-1206(10)62144-8. PMID 12602669
- [Background] Philip G, Malmstrom K, Hampel FC, Weinstein SF, LaForce CF, Ratner PH, Malice MP, Reiss TF; Montelukast Spring Rhinitis Study Group. Montelukast for treating seasonal allergic rhinitis: a randomized, double-blind, placebo-controlled trial performed in the spring. Clin Exp Allergy. 2002 Jul;32(7):1020-8. doi: 10.1046/j.1365-2222.2002.01422.x. PMID 12100048
- [Background] Nayak AS, Philip G, Lu S, Malice MP, Reiss TF; Montelukast Fall Rhinitis Investigator Group. Efficacy and tolerability of montelukast alone or in combination with loratadine in seasonal allergic rhinitis: a multicenter, randomized, double-blind, placebo-controlled trial performed in the fall. Ann Allergy Asthma Immunol. 2002 Jun;88(6):592-600. doi: 10.1016/S1081-1206(10)61891-1. PMID 12086367
- [Background] Pullerits T, Praks L, Ristioja V, Lotvall J. Comparison of a nasal glucocorticoid, antileukotriene, and a combination of antileukotriene and antihistamine in the treatment of seasonal allergic rhinitis. J Allergy Clin Immunol. 2002 Jun;109(6):949-55. doi: 10.1067/mai.2002.124467. PMID 12063523
- [Background] Wilson AM, Sims EJ, Orr LC, Coutie WJ, White PS, Gardiner Q, Lipworth BJ. Effects of topical corticosteroid and combined mediator blockade on domiciliary and laboratory measurements of nasal function in seasonal allergic rhinitis. Ann Allergy Asthma Immunol. 2001 Oct;87(4):344-9. doi: 10.1016/S1081-1206(10)62250-8. PMID 11686428
- [Background] Wilson AM, Dempsey OJ, Sims EJ, Lipworth BJ. A comparison of topical budesonide and oral montelukast in seasonal allergic rhinitis and asthma. Clin Exp Allergy. 2001 Apr;31(4):616-24. doi: 10.1046/j.1365-2222.2001.01088.x. PMID 11359431
- [Background] Wilson AM, Orr LC, Sims EJ, Lipworth BJ. Effects of monotherapy with intra-nasal corticosteroid or combined oral histamine and leukotriene receptor antagonists in seasonal allergic rhinitis. Clin Exp Allergy. 2001 Jan;31(1):61-8. PMID 11167952
- [Background] Wilson AM, Orr LC, Sims EJ, Dempsey OJ, Lipworth BJ. Antiasthmatic effects of mediator blockade versus topical corticosteroids in allergic rhinitis and asthma. Am J Respir Crit Care Med. 2000 Oct;162(4 Pt 1):1297-301. doi: 10.1164/ajrccm.162.4.9912046. PMID 11029334
- [Derived] Esteitie R, deTineo M, Naclerio RM, Baroody FM. Effect of the addition of montelukast to fluticasone propionate for the treatment of perennial allergic rhinitis. Ann Allergy Asthma Immunol. 2010 Aug;105(2):155-61. doi: 10.1016/j.anai.2010.05.017. Epub 2010 Jun 19. PMID 20674827

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were seen at the Nasal Physiology Laboratory at the University of Chicago.
Pre-assignment Details: Those having residual symptoms (total nasal symptom score of 4+) after the open-label phase were randomized to montelukast or placebo for another two weeks in addition to fluticasone propionate. Of the 102 subjects in open-label phase, 54 with residual symptoms were randomized and are listed as "completed" in open-label period of participant flow.
Groups:
- Fluticasone Propionate Only: Fluticasone propionate nasal spray - 2 sprays in each nostril once a day (200 micrograms daily)
- Fluticasone Propionate+Montelukast: Fluticasone propionate nasal spray - 2 sprays in each nostril once a day (200 micrograms daily)
  Montelukast - 10 mg po daily
- Fluticasone Propionate+Placebo: Fluticasone propionate nasal spray - 2 sprays in each nostril once a day (200 micrograms daily)
  Placebo - 10 mg po daily
Period: Open-Label Phase (2 Weeks)
Arm/Group | Fluticasone Propionate Only | Fluticasone Propionate+Montelukast | Fluticasone Propionate+Placebo
Started | 102 | 0 | 0
Completed | 54 | 0 | 0
Not Completed | 48 | 0 | 0
Not completed — Did not have residual symptoms | 48 | 0 | 0
Period: Double-Blind, Randomized Phase (2 Weeks)
Arm/Group | Fluticasone Propionate Only | Fluticasone Propionate+Montelukast | Fluticasone Propionate+Placebo
Started | 0 | 28 (Baseline Analysis Population) | 26 (Baseline Analysis Population)
Completed | 0 | 28 | 26
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluticasone Propionate + Montelukast | Fluticasone Propionate + Placebo | Total
Number analyzed (Participants) | 28 | 26 | 54
Age, Continuous [Mean (Full Range); unit: years] | 35 [19 to 56] | 32 [18 to 52] | 34 [18 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 15 | 35
  Male | 8 | 11 | 19
Race/Ethnicity, Customized [Number; unit: participants]
  White | 11 | 13 | 24
  Black or African American | 16 | 11 | 27
  Hispanic | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 28 | 26 | 54

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Nasal Symptom Score (TNSS) Over 2 Week Randomized Treatment Period
Description: Patients recorded the severity of sneezing, runny nose, stuffy nose, and other symptoms (itchy nose/eyes and post-nasal drip) twice a day on a scale from 0 to 3 (0 = no symptoms, 1 = mild, 2 = moderate, and 3 = severe). The TNSS was calculated as the sum of all scores for morning and evening recordings with a range of 0 to 24.
  The baseline TNSS used in the analysis was the average of the symptom scores from the last 5 days of fluticasone propionate therapy prior to randomized treatment period.
  The change from baseline for each subsequent day of treatment was then calculated for each subject. So that each subject only had one observation, the average of these changes was calculated for each subject, and this summary measure was used in the analysis comparing the two treatment groups. We report the median and full range of these average changes for each group.
  A negative value indicates an improvement in symptoms.
Time Frame: Baseline and 2 weeks
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Fluticasone Propionate + Montelukast | Fluticasone Propionate + Placebo
Number analyzed (Participants) | 28 | 26
units on a scale | -1.66 [-17.85 to 1.69] | -2.21 [-13.82 to 4.5]
Statistical Analysis 1: Comparison: Fluticasone Propionate + Montelukast vs Fluticasone Propionate + Placebo; Test type: Superiority or Other; p = 0.8, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change From Baseline in Sneezing Symptom Score Over 2 Week Randomized Treatment Period
Description: Patients recorded the severity of sneezing twice a day on a scale from 0 to 3 (0 = no symptoms, 1 = mild, 2 = moderate, and 3 = severe). The sneezing symptom score was calculated as the sum of all scores for morning and evening recordings with a range of 0 to 6.
  The baseline symptom score used in the analysis was the average of the symptom scores from the last 5 days of fluticasone propionate therapy prior to randomized treatment period.
  The change from baseline for each subsequent day of treatment was then calculated for each subject. So that each subject only had one observation, the average of these changes was calculated for each subject, and this summary measure was used in the analysis comparing the two treatment groups. We report the median and full range of these average changes for each group.
  A negative value indicates an improvement in symptoms.
Time Frame: Baseline and 2 weeks
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Fluticasone Propionate + Montelukast | Fluticasone Propionate + Placebo
Number analyzed (Participants) | 28 | 26
units on a scale | -0.22 [-5.62 to 2.0] | -0.25 [-2.57 to 2.68]
Statistical Analysis 1: Comparison: Fluticasone Propionate + Montelukast vs Fluticasone Propionate + Placebo; Test type: Superiority or Other; p = 0.70, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change From Baseline in Runny Nose Symptom Score Over 2 Week Randomized Treatment Period
Description: Patients recorded the severity of runny nose twice a day on a scale from 0 to 3 (0 = no symptoms, 1 = mild, 2 = moderate, and 3 = severe). The runny nose symptom score was calculated as the sum of all scores for morning and evening recordings with a range of 0 to 6.
  The baseline symptom score used in the analysis was the average of the symptom scores from the last 5 days of fluticasone propionate therapy prior to randomized treatment period.
  The change from baseline for each subsequent day of treatment was then calculated for each subject. So that each subject only had one observation, the average of these changes was calculated for each subject, and this summary measure was used in the analysis comparing the two treatment groups. We report the median and full range of these average changes for each group.
  A negative value indicates an improvement in symptoms.
Time Frame: Baseline and 2 weeks
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Fluticasone Propionate + Montelukast | Fluticasone Propionate + Placebo
Number analyzed (Participants) | 28 | 26
units on a scale | -0.52 [-3.85 to 1.08] | -0.29 [-2.60 to 2.42]
Statistical Analysis 1: Comparison: Fluticasone Propionate + Montelukast vs Fluticasone Propionate + Placebo; Test type: Superiority or Other; p = 0.86, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change From Baseline in Stuffy Nose Symptom Score Over 2 Week Randomized Treatment Period
Description: Patients recorded the severity of stuffy nose twice a day on a scale from 0 to 3 (0 = no symptoms, 1 = mild, 2 = moderate, and 3 = severe). The stuffy nose symptom score was calculated as the sum of all scores for morning and evening recordings with a range of 0 to 6.
  The baseline symptom score used in the analysis was the average of the symptom scores from the last 5 days of fluticasone propionate therapy prior to randomized treatment period.
  The change from baseline for each subsequent day of treatment was then calculated for each subject. So that each subject only had one observation, the average of these changes was calculated for each subject, and this summary measure was used in the analysis comparing the two treatment groups. We report the median and full range of these average changes for each group.
  A negative value indicates an improvement in symptoms.
Time Frame: Baseline and 2 weeks
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Fluticasone Propionate + Montelukast | Fluticasone Propionate + Placebo
Number analyzed (Participants) | 28 | 26
units on a scale | -0.41 [-5.31 to 2.37] | -0.47 [-4.53 to 2]
Statistical Analysis 1: Comparison: Fluticasone Propionate + Montelukast vs Fluticasone Propionate + Placebo; Test type: Superiority or Other; p = 0.48, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change From Baseline in Other Symptom Score Over 2 Week Randomized Treatment Period
Description: Patients recorded the severity of other symptoms, including itchy nose/eyes and post-nasal drip, twice a day on a scale from 0 to 3 (0 = no symptoms, 1 = mild, 2 = moderate, and 3 = severe). The other symptom score was calculated as the sum of all scores for morning and evening recordings with a range of 0 to 6.
  The baseline symptom score used in the analysis was the average of the symptom scores from the last 5 days of fluticasone propionate therapy prior to randomized treatment period.
  The change from baseline for each subsequent day of treatment was then calculated for each subject. So that each subject only had one observation, the average of these changes was calculated for each subject, and this summary measure was used in the analysis comparing the two treatment groups. We report the median and full range of these average changes for each group.
  A negative value indicates an improvement in symptoms.
Time Frame: Baseline and 2 weeks
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Fluticasone Propionate + Montelukast | Fluticasone Propionate + Placebo
Number analyzed (Participants) | 28 | 26
units on a scale | -0.24 [-3.40 to 1.25] | -0.14 [-4.35 to 1.22]
Statistical Analysis 1: Comparison: Fluticasone Propionate + Montelukast vs Fluticasone Propionate + Placebo; Test type: Superiority or Other; p > 0.99, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: During the two weeks of randomized treatment
Arm/Group | Fluticasone Propionate + Montelukast | Fluticasone Propionate + Placebo
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/26
Other Adverse Events (participants affected / at risk) | 0/28 | 0/26

LIMITATIONS AND CAVEATS:
Early termination of study due to difficulty recruiting

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No